CLINICAL TRIAL: NCT01917864
Title: Handheld Technology for Speech Development in Students With Autism Spectrum Disorders
Brief Title: iPad Application to Treat Prosodic Deficits in Students With Communication Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Handhold Adaptive (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1306012259; ED-IES-13-R-0005 (Other Grant/Funding Number: Department of Education)
Record Dates: First submitted 2013-08-05; First posted 2013-08-07 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Autism; Communication Disorders
Keywords: Autism; Autism Spectrum Disorders; Prosody; Speech treatment
MeSH Terms: conditions — Autistic Disorder; Communication Disorders; Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- iPad Application (Experimental): Student participants will use specialized iPad software under the supervision of a speech-language pathologist over the course of 12 months, approximately one session per week, one hour per session.
  Interventions: Behavioral: iPad Application

INTERVENTIONS:
Behavioral: iPad Application — A specialized iPad application, entitled SpeechPrompts, has been developed to treat prosodic difficulties commonly seen in ASDs. SpeechPrompts provides the SLPs that work with students with ASDs an additional tool to treat prosody. The SpeechPrompts software offers visual support and biofeedback to change prosody. These two tools are not typically available for school-based SLPs.

SUMMARY:
The purpose of this study is to evaluate the utility of a specialized iPad application designed to treat difficulties with intonation (e.g., melody in voice) in children with autism spectrum disorders (ASD) and other communication disorders.

ELIGIBILITY:
Inclusion Criteria:

* SLPs, in Connecticut Public Schools, who provide intervention to students with autism spectrum disorders and related disorders
* Students, ages 4-18, who attend school in Connecticut and demonstrate prosodic difficulties secondary to a diagnosis of ASD, apraxia of speech, or other communication disorder

Exclusion Criteria:

* Students with concomitant genetic disorders

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-07; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Effectiveness of software | 12 months
  The effectiveness of the software will be measured in two ways.
  1. Perceptual ratings of prosody. Pre- and post-treatment speech samples will be collected from each student participant. These samples will be rated by a member of the research staff on the following prosodic characteristics: rate, rhythm, stress, volume.
  2. Questionnaires. Questionnaires will be completed pre- and post-treatment by the students' classroom teacher and speech-language pathologist. These questionnaires will measure the students' use and generalization of skills taught during the intervention.

SECONDARY OUTCOMES:
Usability of software | 12 months
  Usability of software will be measured through questionnaires completed by the speech-language pathologists. Questionnaires will measure ease of software use, utility of software functions, and student engagement during intervention sessions.
Student engagement in treatment | 12 months
  Student engagement will be evaluated indirectly by rating scales completed by the speech-language pathologist. Likert scales will be used to quantify student engagement on the following parameters: time engaged in on-task behavior, time engaged in off-task behavior, perceived enjoyment of software.
Improvement in peer acceptance | 12 months
  Changes in peer acceptance will be evaluated using two different methodologies.
  1. Classroom teacher questionnaire. Each student's classroom teacher will complete a questionnaire pre- and post-treatment measuring the student's interaction with classroom peers.
  2. Semi-structured observation. A member of the research staff will observe each student pre- and post-treatment and complete frequency tallies on the number of peer interactions initiated during a 15-minute semi-structured activity.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Shic, Ph.D, Principal Investigator — Yale University
Locations (1):
- Yale Child Study Center, New Haven, Connecticut, United States